CLINICAL TRIAL: NCT06441994
Title: A Phase I Investigator-initiated Clinical Trial of a Novel Targeted Alpha Therapy Using [At-211]PSMA-5 for Patients With Castration-resistant Prostate Cancer
Brief Title: Clinical Trial of Targeted Alpha Therapy Using [At-211]PSMA-5 for Prostate Cancer
Acronym: Alpha-PS1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Osaka University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Tadashi Watabe, Associate Professor, Osaka University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APS1-001
Record Dates: First submitted 2024-05-26; First posted 2024-06-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Astatine (At-211); Targeted alpha therapy; PSMA (Prostate Specific Membrane Antigen)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration arm (Experimental)
  Interventions: Drug: PSW-1025

INTERVENTIONS:
Drug: PSW-1025 — PSMA (prostate specific membrane antigen)-targeted alpha therapy drug labeled with Astatine (At-211)

SUMMARY:
PSW-1025 is administered intravenously to patients with castration-resistant prostate cancer to evaluate its tolerability, safety, pharmacokinetics, absorbed dose, and efficacy, as well as to determine the recommended dose for Phase II.

DETAILED DESCRIPTION:
PSW-1025 is administered intravenously to patients with castration-resistant prostate cancer to evaluate its tolerability, safety, pharmacokinetics, absorbed dose, and efficacy, as well as to determine the recommended dose for Phase II. PSW-1025 ([At-211]PSMA-5) is an alpha-ray-emitting drug labeled with Astatine (At-211) that targets PSMA (Prostate Specific Membrane Antigen).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with progressive castration-resistant prostate cancer who meet the following conditions (1) and (2) (1) Patients with progressive increase of serum Prostate-Specific Antigen (PSA) (>=2ng/mL, three consecutive increases at least one week apart, and two increases of more than 50% from the lowest value), or with the tumor growth or appearance of new lesions detected by imaging studies (2) Patients with the serum testosterone at castration level (< 50ng/dL)
2. Patients who meet the following conditions (1) and (2), resistant to standard treatment or not indicated for the generally approved standard treatments (1) Patients who have received at least one of the following treatments

   * Inhibitors of androgen receptor signaling (enzalutamide, apalutamide, dalortamide, etc.)
   * Inhibitors of Cytochrome P450 17 (CYP 17) (abiraterone acetate) (2) Patients previously treated with the taxane-based chemotherapy (docetaxel or cabazitaxel) or not adapted for the taxane-based chemotherapy (including refusal cases)* * Targeting for the patients who have received cabazitaxel therapy after docetaxel therapy, or patients for whom cabazitaxel therapy was not indicated (including refusal cases) after docetaxel therapy, or patients for whom both docetaxel therapy and cabazitaxel therapy were not indicated (including refusal cases)
3. Patients aged 18 years or older at the time of consent acquisition
4. Patients with stable general condition with PS (Performance status) of 0 to 2 in ECOG (Eastern Cooperative Oncology Group)
5. Patients who can be expected to survive for 6 months or more, judging from clinical symptoms and medical examination findings
6. Patients without or with controlled symptomatic brain metastases
7. Patients with no clinically significant abnormal findings in electrocardiogram, respiratory rate, and blood oxygen saturation within 30 days before the enrollment
8. Patients whose laboratory values within 30 days before the enrollment are within the range specified in the protocol
9. Patients who can use appropriate contraception during the clinical trial period according to the protocol
10. Patients who thoroughly listened to the explanation of the clinical trial, agreed to the various study procedures outlined in the clinical trial protocol and signed the consent document

Exclusion Criteria:

1. Patients who received systemic antitumor therapy (e.g. chemotherapy, immunotherapy, biologic therapy such as monoclonal antibodies, excluding androgen receptor signaling inhibitors) within 4 weeks before enrollment
2. Patients who received radium chloride (Radium, 223Ra) or 177Lu (Lutetium)-PSMA-617 within 6 months before registration
3. Patients currently receiving treatment with other cytotoxic chemotherapy, immunotherapy, radioligand therapy, poly adenosine diphosphate-ribose polymerase (PARP) inhibitors, AKT inhibitors
4. Patients with active double cancer (simultaneous double cancer and ectopic double cancer with a disease-free period of 5 years or less)
5. Patients who received other investigational drugs within 5 weeks prior to enrollment
6. Patients with uncontrollable active infections
7. Hepatitis B surface antigen positive, Hepatitis C Virus antibody positive (patients with HCV-RNA level below the limit of detection can be registered) or Human Immunodeficiency Virus antibody positive patients
8. Patients with mental illness or psychiatric symptoms who are judged to be difficult to participate in clinical trials
9. Other patients who are judged to be inappropriate by the investigator, etc.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events as assessed by CTCAE v5.0 | until 6 months after administration
Dose Limiting Toxicity | within 4 weeks after single administration

SECONDARY OUTCOMES:
Number of participants with adverse events and their details | until 6 months after administration
Blood pressure (mmHg) and heart rate (bpm) | until 6 months after administration
Symptoms of the participants | until 6 months after administration
Hematological tests (blood cell counts) | until 6 months after administration
Urine tests (occult blood and urine protein) | until 6 months after administration
Electrocorticogram | until 6 months after administration
Prostate-Specific Antigen (PSA) (ng/ml) | until 6 months after administration
Tumor size on CT (mm) | until 6 months after administration
Excretion rates in urine, feces, and breath (%injected dose) | until 24 hours after administration
Absorbed doses in major organs (Gy) | until 24 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No